CLINICAL TRIAL: NCT02317614
Title: SteadyRx: Smartphone ART Adherence Intervention for Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00026315; R34DA037130 (NIH)
Record Dates: First submitted 2014-12-10; First posted 2014-12-16 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: HIV; Medication Adherence
Keywords: Incentives; Smartphone; Mobile intervention; eDOT; Adherence reinforcement; Drug users
MeSH Terms: conditions — Medication Adherence; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SteadyRx (Experimental): This group will be assessed at monthly intervals. They will receive their usual care at their regular providers. In addition, they will be given Smartphones loaded with the SteadyRx intervention.
  Interventions: Behavioral: SteadyRx
- Usual Care (No Intervention): This group will be assessed at monthly intervals. They will receive their usual care at their regular providers. They will not receive a Smartphone or the SteadyRx adherence intervention.

INTERVENTIONS:
Behavioral: SteadyRx — The proposed intervention consists of four core elements. The intervention will include a Smartphone application that allows direct interaction with the SteadyRx system, as well as automatic events controlled via a central server. The CONSULT element will facilitate patient-provider communication with links to care providers and other care resources. The REMIND element will provide telephonic reminders for late doses. The OBSERVE element will feature electronically observed dosing through time-stamped video recordings made on the Smartphone and sent securely to a central server. The REWARD element will feature monetary incentives designed to reinforce short- and long-term medication adherence and promote reductions in viral load.
  Arms: SteadyRx

SUMMARY:
Antiretroviral therapy (ART) increases life expectancy and quality of life for individuals infected with HIV, and can reduce the chance of HIV transmission, but a high degree of adherence to ART is required to achieve these benefits. Unfortunately, only 59% of patients in North America report ART adherence >90%. Thus, ART adherence interventions are a critical part of the fight against HIV/AIDS. Injection drug use and crack cocaine use are major factors in the transmission of HIV, and are associated with non-adherence to ART. Several types of interventions, most notably directly administered antiretroviral therapy (direct observation of antiretroviral administration and patient supports) and contingency management (the provision of incentives contingent upon objective evidence of adherence) have been effective in promoting ART adherence in drug users. However, a core problem with all ART adherence interventions is that their effects do not last after the interventions are discontinued. The common finding of post-intervention dissipation of effects suggests that ART adherence interventions may need to be long-term or even permanent adjuncts to ART for drug users. The investigators intend to develop an intensive intervention that incorporates the most effective techniques for promoting ART adherence in drug users, and delivers them in a manner that allows for their large-scale implementation as long-term or even permanent adjuncts to ART. Thus, we will bundle a targeted group of effective component interventions into a smartphone application that is easy for patients to use, simple to manage, and maximally convenient for all stakeholders. Our ultimate goal is to produce an intervention that is highly effective and scalable. Toward that end, the SteadyRX intervention to be developed under this project will be largely automated and will (1) facilitate consultation with care providers (2) provide reminders when a dose is overdue, (3) provide electronic remote observation of medication-taking, and (4) reward ART adherence. In addition to developing this smartphone-based intervention, a pilot study will be conducted in 50 HIV+ adults with a history of problem drug use. In this study, participants will be randomly assigned to receive usual care, or usual care plus the SteadyRX intervention.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) increases life expectancy and quality of life for individuals infected with HIV, and can reduce the chance of HIV transmission. These fantastic personal and public health benefits require a high level of adherence to the prescribed treatment regimen. High rates of virologic suppression can be achieved with an adherence rate of 90%, but adherence of 95% or more appears to produce the best combination of a higher probability of virologic suppression and a lower probability of the development of resistance to the medications. Unfortunately, only 59% of patients in North America report ART adherence >90%. Thus, ART adherence interventions are a critical part of the fight against HIV/AIDS, and there is a substantial need for novel and effective ART adherence interventions.

Injection drug use and crack cocaine use are major factors in the transmission of HIV and have been associated with non-adherence to ART. Several types of interventions have been effective in promoting short-term ART adherence in these populations. Counseling strategies and reminders (e.g., beepers, calendars, etc.) have each had modest effects. Still more successful approaches have included directly administered antiretroviral therapy (DAART, in which patients are observed by care providers as they take their medication), medication assisted therapy (e.g., methadone maintenance), and contingency management (monetary incentives for maintaining adherence to HIV medications). However, a core problem with all ART adherence interventions is that their effects do not appear to last after the interventions are discontinued. In a recent review of ART adherence interventions for drug users, researchers expressed concern over the "virtual lack of interventions with sustained post-intervention adherence and virologic benefits." The common finding of post-intervention dissipation of effects suggests that ART adherence interventions may need to be implemented as long-term or even permanent adjuncts to ART for drug users.

The investigators seek to develop an intensive intervention that incorporates the most effective techniques for promoting ART adherence in drug users, and deliver them in a manner that allows for their large-scale implementation as long-term or even permanent adjuncts to ART. The investigators propose a three year development project for an ART adherence intervention that bundles a targeted group of effective component interventions into a Smartphone application that is easy for patients to use, simple to manage, and maximally convenient for all stakeholders. Toward that end, the intervention to be developed under this project will (1) facilitate consultation with care providers (2) provide reminders when a dose is overdue, (3) provide remote electronic observation of medication-taking, and (4) provide incentives for ART adherence. The proposed intervention (SteadyRx) is highly innovative: no previous ART adherence intervention has involved direct observation of medication administration and contingency management, despite their respective effectiveness in isolation. Importantly, no mobile/remote intervention currently under development is as intensive as SteadyRx.

The developmental process for this application will begin with modification of existing technology, which will be followed by conducting focus groups with the intended target population as well as with physicians, primary care staff, and health administrators, respectively, in order to enhance the adoptability of the intervention by including application functions and interface design that is sensitive to the needs of all stakeholders. Small scale testing with members of the target population will be used to further refine the application and produce a beta version for use in a pilot randomized controlled trial.

In the pilot study, 50 HIV+ adults with a history of problem drug use will be randomly assigned to receive either usual care services at a primary care facility or these services plus the SteadyRx intervention. The project has the following Specific Aims:

1. Develop the SteadyRx Smartphone intervention

   1. Conduct focus groups with the target population, physicians, primary care staff, and health administrators, respectively, prior to creating the application and instructional materials
   2. Create alpha versions of the smartphone application and related instructional materials
   3. Create a beta version of the application to use in the pilot randomized controlled trial.
2. Implement SteadyRx in a pilot randomized controlled trial

   1. Evaluate SteadyRx's acceptability to stakeholders, user experience, and user engagement.
   2. Collect preliminary data on the effectiveness of SteadyRx in improving ART adherence, reducing viral load, and promoting high CD4 counts
   3. Collect preliminary assessment of associations between ongoing drug use and health literacy and the effectiveness of SteadyRx.

Overall, the combination of consultation, reminders, direct observation, and incentives for adherence, when delivered as a long-term adjunct to ART via Smartphone application could prove to be a maximally effective and practical means of realizing the fantastic potential of modern ART for improving the lives of individuals with HIV/AIDS and for reducing the rate of HIV transmission by high-risk patients.

STUDY PROCEDURES Application Development Alpha Version. As the first step in the development of the application, the investigators will create an alpha version of the application that includes the PillWatch feature. Note that the PillWatch feature will require only minor modification from the existing Mōtiv8 technology used by Dallery (Co-I). Other aspects of the planned application will require more substantial development and thus will not be fully developed until after the focus group sessions described below.

Focus Groups. As the second step in the development of the application, the investigators will conduct three focus group sessions. All focus groups will be designed and moderated by Baltimore Research, a full service marketing research company with over 50 years of experience (See Facilities and Other Resources for further details). Baltimore Research will also handle all data collection and analysis for the focus group sessions and provide the study team with a final report for each session. Each focus group will include a relatively homogeneous set of stakeholders: Physicians/primary care staff, health administrators (e.g., see Priority Partners letter of support), and patients, respectively. All focus groups will include approximately eight participants, as this has been identified as an ideal number of participants in a focus group session. In order to ensure that approximately eight participants will be included, the investigators will attempt to recruit at least 10 participants, because all participants must show up at the same time for a specific scheduled session, and this usually results in some people who agree to participate but do not show up at the scheduled time. These groups will be held as one-time sessions designed to generate ideas that will enhance the application's usability and adoptability from the perspective of the professionals who are most likely to be involved in the institutional decision making processes relevant to the dissemination of the proposed intervention. The investigators anticipate that recruitment of health professionals will be straightforward given our extensive connections to professionals throughout the local health care systems in Baltimore, and consultation by Baltimore Research will ensure that these recruitment processes are free of bias. The third focus group session (patients) will be the beginning of an iterative process in which the investigators first solicit ideas about the functionality and interface of the application. Participants for this focus group will be recruited using methods identical to those described below for the pilot randomized controlled trial.

Create the Beta Version. Following the initial four focus group sessions, the beta version of the application will be created with the critical features described above. The end product of this part of the development process will be the beta version that will be used in the pilot study described below.

PILOT STUDY The investigators expect that all participants will be patients at the Comprehensive Care Practice (CCP). CCP is located in the Mason F. Lord Building at the Johns Hopkins Bayview Medical Center in Baltimore, MD. CCP provides primary medical care to ~450 HIV+ adults and will serve as the recruitment site.

Participants will be recruited from their regularly scheduled HIV care appointments at the CCP at which current viral load and CD4 counts are evaluated. Any HIV+ patient with a substance use disorder will be told by their CCP doctor about our research study and given a recruitment flyer that explains the benefits of participation. If they express interest, the doctor will immediately contact the CCP Medical Case Manager who is in charge of study recruitment and assessment (hereafter, outreach coordinator). The outreach coordinator will briefly explain the intake interview process and basic purpose of the study. If the patient agrees to move forward they will begin with a formal consent process. During this process, the outreach coordinator will read the consent form aloud in its entirety while the participant follows along. After signing the consent form, the patient will proceed immediately to the intake interview unless their schedule precludes it, in which case they will provide contact information and schedule the intake interview for a time on the next day or as soon as possible. Participants who have signed consent but who have not returned to CCP will be given reminder calls related to their scheduled intake interview. They will also receive follow up calls if they fail to show up for their scheduled appointment time.

For any given pilot study participant, study participation will last for six months, and will include an intake visit plus six visits at 30 day intervals thereafter. For focus group participants, study participation will consist of a single focus group session.

ELIGIBILITY:
Inclusion Criteria:

* Applicants will be eligible to participate in the study if they:

  1. are 18 to 100 years old;
  2. are HIV positive;
  3. have a primary care physician who is providing their HIV-related care including prescribed ART;
  4. have a substance use disorder
  5. can operate a smartphone
  6. speak English fluently

Exclusion Criteria:

* Applicants will be excluded if they:

  1. report current suicidal or homicidal ideation;
  2. report active hallucinations;
  3. are participating in another HIV related study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fingerhood, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Comprehensive Care Practice, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The originally planned recruitment strategy did not work. We thus expanded our recruitment to the entire city of Baltimore instead of just one clinic.
Period: Overall Study
Arm/Group | SteadyRx | Usual Care
Started | 26 | 25
Completed (1 non-complete lost to follow-up prior to accessing intervention (immediately after enrollment)) | 23 | 23
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: The participant who was lost to follow-up immediately after study enrollment is not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | SteadyRx | Usual Care | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.36 (10.69) | 54 (7.81) | 53.18 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 8 | 16 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 23 | 21 | 44
  White | 1 | 3 | 4
  Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Education (years) [Mean (Standard Deviation); unit: years] | 11.96 (1.24) | 11.88 (2.13) | 11.92 (1.69)
Test of Functional Health Literacy in Adults (TOFHLA) score [Mean (Standard Deviation); unit: units on a scale] — The TOFHLA has two main sections, one for reading literacy and one for numeracy. These are each scored from zero to 50 then summed for a composite score. Composite scores less than 60 indicate inadequate health literacy. Scores between 60 and 74 indicate marginal health literacy. Scores 75 and above indicate adequate health literacy.
  units on a scale | 85.16 (12.36) | 80.28 (15.27) | 82.72 (13.82)
number (and percentage) of participants with clinical depression [Count of Participants; unit: Participants] | 9 | 11 | 20
number (and percentage) of participants with cocaine or non-prescribed opioids in the last 30 days [Count of Participants; unit: Participants] | 9 | 6 | 15
number (and percentage) of participants with cocaine or non-prescribed opioid use in their lifetime [Count of Participants; unit: Participants] | 24 | 23 | 47
number (and percentage) of participants with an undetectable HIV viral load [Count of Participants; unit: Participants] | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence as Assessed by the Medication Event Monitoring System (MEMS) Cap
Description: The MEMS cap is a device that records the date and time whenever a patient opens a vial to monitor medication adherence. Percentage of participant to achieve 95% adherence will then be recorded.
Time Frame: Six months
Population: Participants' monthly data over six months were included. Missing data were treated as missing.
Measure: Number; unit: percentage of participants
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
percentage of participants | 52.2 | 27.2

2. Primary Outcome: Percentage of Participants Achieving an Undetectable Viral Load in Six Months
Description: Measured twice in six months to assess the percentage of participants to achieve a viral load <400 HIV-RNA/mL (Y/N)
Time Frame: Six months
Measure: Number; unit: percentage of participants
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
percentage of participants | 88.1 | 100

3. Secondary Outcome: Monthly Percent Adherence to Antiretroviral Medications.
Description: This measure is calculated for each participant in each study month. The number of days in the month in which the participant correctly consumed their antiretroviral medication is divided by the number of days in the month. The measure is collected by an electronic pill bottle cap (a.k.a. "MEMS cap").
Time Frame: Six months
Measure: Mean (Standard Error); unit: percentage of adherence to ART
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
percentage of adherence to ART | 87.97 (1.64) | 73.88 (2.4)

4. Secondary Outcome: Viral Load
Description: Actual HIV-RNA levels, measured at the same time as the undetectable viral load outcome measure
Time Frame: Six months
Measure: Mean (Standard Error); unit: copies/mL blood
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
copies/mL blood | 248.17 (182.64) | 23.38 (1.37)

5. Other Pre Specified Outcome: Mental and Physicial Health as Assessed by the Medical Outcomes Study HIV Health Survey (MOS-HIV)
Description: The 35-item questionnaire includes ten dimensions (health perceptions, pain, physical, role, social and cognitive functioning, mental health, energy, health distress and quality of life (QoL). Subscales are scored on a 0-100 scale (a higher score indicates better health) and separate physical and mental health summary scores are calculated. Summary scores for these items are transforms with a mean of 50 and a standard deviation of 10. Thus, for both scores, being of average (physical or mental) health leads to a score of 50, with a range of 20 to 80.
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Mental health score | 54.6 (8.33) | 51.4 (12.36)
  Physical health score | 45.63 (11.41) | 42.75 (12.95)

6. Other Pre Specified Outcome: Opiate and Cocaine Use
Description: Measured using monthly self-report. Response will be binary (Yes/No). The percentage of the participants that reported yes will be recorded for each month and then an average for the 6 month period calculated.
Time Frame: Six months
Population: Includes data from six months (repeated measures), with missing data treated as missing. Percent of participants reporting use of either cocaine, opiates, or both is the reported value.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | SteadyRx | Usual Care
Number analyzed (Participants) | 25 | 25
percentage of participants | 20.0 (9.0) | 22.8 (4.9)

ADVERSE EVENTS:
Time Frame: 6 months
Description: The FDA definition of adverse events was used to guide adverse event reporting to the funding agency and IRB during this study. According to the FDA definition, no adverse events occurred during the monitoring period. In addition, adverse events were recorded based on the clinicaltrials.gov definitions.
Arm/Group | SteadyRx | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SteadyRx (N=25) | Usual Care (N=25)
Death (Immune system disorders) | 1 (1) | 1 (1)
Hospitalization (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02317614/Prot_SAP_000.pdf